CLINICAL TRIAL: NCT04822428
Title: Effect of Visceral Osteopathic Manipulations on Low Back Pain Caused by Visceral Dysfunctions
Brief Title: Effect of Visceral Osteopathic Manipulations on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SH2021
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, parallel study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group(A) (Experimental): Group (A): included Twenty patients who received osteopathic manipulative techniques, 1 session per week for 3 weeks.
  Interventions: Other: Osteopathic manipulation
- Control group(B) (No Intervention): Group (B): included twenty patients who received analgesic drugs only.

INTERVENTIONS:
Other: Osteopathic manipulation — Osteopathic manipulative techniques including; suboccipital release technique,sacral release technique, diaphragmatic release, mesentery release, and Colonic manipulation
  Arms: study group(A)

SUMMARY:
Forty female patients with age ranging from 30-40 years old were suffering from low back pain due to visceral dysfunctions participated in this study. They were recruited from a private clinic. They were assigned into two groups equal in number; Group (A): included twenty patients who received osteopathic manipulative techniques, 1 session per week for 3 weeks, and Group (B): included twenty patients who received only analgesic drugs.

DETAILED DESCRIPTION:
Twenty patients received osteopathic manipulative techniques including Suboccipital release technique, diaphragmatic release.,mesentery release and Colonic manipulation were applied to the study group according to the patients' needs.

The treatment program comprised a total of 3 sessions for 3 weeks at one session per week for an average of 50 minutes per session. Twenty patients in the second group (control ) took only analgesics during the three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain for more than 12 weeks

Exclusion Criteria:

* Malignant tumor
* Pregnancy
* Acute ischemic bowel disease,
* Intestinal obstruction,
* surgery in the last six months

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
The visual analog scale (VAS) | change from baseline to after 3 weeks
  The patient determined the pain intensity on a 10 cm scale marked with points ranging from predetermined no pain and excruciating pain
The Oswestry Disability Index (ODI) | change from baseline to after 3 weeks
  (ODI) consists of 10 items on the degree of severity to which back (or leg) trouble has affected the ability to manage in everyday life.
Modified Schober's test (MST) | change from baseline to after 3 weeks
  the participant stood erect while the lumbosacral junction was marked as indicated by the dimples of Venus. For measuring the MST, we put a mark 5 cm below and 10 cm above the junction. The participant was asked to bend forward as far as possible and the stretched distance of these two points was measured as the MST value.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No